CLINICAL TRIAL: NCT02037490
Title: Grow2Gether: Pilot Trial of a Peer-Based Social Media Intervention to Promote Healthy Growth During Infancy
Brief Title: Grow2Gether Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-010702
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Childhood Obesity
Keywords: Infants; Mothers; Social media; Obesity prevention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grow2Gether Intervention (Experimental): Participants in the intervention group will:
  * Participate in the Grow2Gether intervention
  * Receive text message reminders, 1) to schedule recommended primary care visits for their infant, and 2) to attend appointments scheduled in CHOP Care Network.
  Interventions: Behavioral: Grow2Gether
- Control (No Intervention): Participants in the control group will:
  * Receive text message reminders, 1) to schedule recommended primary care visits for their infant, and 2) to attend appointments scheduled in CHOP Care Network.

INTERVENTIONS:
Behavioral: Grow2Gether — Participants in this intervention will:
  Participate in Facebook group of 6-12 peers for about 8 months, led by a professional group mentor.
  Complete an intervention video activity approximately weekly:
  1. View educational videos addressing topics related to healthy infant growth
  2. Create photos/videos modeling healthy behaviors and post them to the group
  3. Provide and receive feedback on posts
  4. Be encouraged to share information with key caregivers of their child
  Attend group party soon after enrollment, to meet peers and group leader in person.
  Arms: Grow2Gether Intervention

SUMMARY:
This is a randomized controlled pilot trial of a peer-based, social media intervention to prevent obesity in infants.

DETAILED DESCRIPTION:
This novel intervention, delivered to mothers primarily through private Facebook groups, will promote behavior change through peer and self-modeling photo/video activities.

In this study, investigators will implement the intervention with small peer groups of 6-12 mothers, beginning during the 3rd trimester of pregnancy. Investigators will assess feasibility and acceptability of the intervention, and explore its impact on outcomes, particularly behaviors associated with healthy growth.

ELIGIBILITY:
Inclusion Criteria:

* Receiving prenatal care from Hospital of the University of Pennsylvania (HUP) obstetrics practices
* Age 18 years and older
* Able to provide informed consent
* Able to speak, read and write in English
* Enrolled in Medicaid at the time of study enrollment
* Overweight or obese (BMI ≥ 25, calculated using height and weight recorded at a prenatal visit prior to 14 weeks of pregnancy)
* In ≥ 20th week of pregnancy
* Plan to receive their child's primary care services from Children's Hospital of Philadelphia (CHOP) Care Network
* Own a smartphone with both a data and text plan
* Able to use their phone to obtain photographs and videos prior to enrollment

Exclusion Criteria:

* Current diagnosis or history of major mental illness, as indicated in medical record by notation of (1) diagnosis or history of condition (2) current use or history of antidepressants or other psychotropic medication, or (3) referral to, or under care of a psychiatrist.
* Multiple pregnancy (twins, triplets, etc.)
* Severe morbidity (significant cardiac disease, significant organ dysfunction, transplant recipient, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability Survey | After (within 31 days of) the 25th/final week of the postnatal intervention curriculum. (Approximately 8 months from each peer group's start.)
  Satisfaction with the overall intervention will be assessed for mothers using a standard survey. Subjects will be asked a series of open-ended and Likert-scaled questions. Additionally, participants with certain characteristics (such as relatively high or low rates of group participation) will be purposively selected for brief semi-structured interviews based on the survey content to further elucidate their opinion of the intervention.
Study population eligibility and interest | At enrollment
  * Proportion of all mothers contacted who meet enrollment criteria
  * Proportion of mothers meeting enrollment criteria who enroll
  These proportions will be calculated using study recruitment records.
Participant engagement | Ongoing with study activities; to be completed after (within 31 days of) the 25th/final week of the postnatal intervention curriculum.
  * Proportion of enrolled mother-infant dyads that comply with intervention participation requirements
  * Proportion of enrolled mother-infant dyads that complete each weekly module activity
  * Proportion of enrolled mother-infant dyads that complete each study measure
  * Number and type of each participant's Facebook group interactions per week (posts, comments, "Likes")
  * Frequency, type, and content of each contact between moderator/study staff and each participant
  This study process data will be obtained from the Facebook group and study records at study end.

OTHER OUTCOMES:
Infant feeding practices | At (or within 31 days of) the infant's newborn primary care visit, and during (or within 31 days of ) the 8th, 17th, and 25th/final week of the postnatal intervention curriculum. (Approx. 2, 4, 6 and 8 months from each peer group's start, respectively.)
  Maternal behaviors related to infant feeding will be measured using 10 items on the Infant Feeding Style Questionnaire (IFSQ). Behavior items are coded on a 5-point scale (never, seldom, half of the time, most of the time, always).
  Also, four items from the validated Infant Feeding Practices Questionnaire (IFPQ) will be used to assess maternal feeding practices related to obesity. The IFPQ contains 20 items, with a 5-point adapted Likert response scale ranging from 0 (Never) to 4 (Always).
Infant feeding beliefs | At (or within 31 days of) the infant's newborn primary care visit, and during (or within 31 days of ) the 25th/final week of the postnatal intervention curriculum. (Approx. 2 and 8 months from each peer group's start, respectively.)
  Maternal beliefs regarding infant feeding will be measured using the Infant Feeding Style Questionnaire (IFSQ), which contains 10 items measuring beliefs, coded on a 5-point scale (disagree, slightly disagree, neutral, slightly agree, agree).
Breastfeeding survey | At enrollment, at (w/in 31 days of) infant's newborn primary care visit, during (w/in 31 days of) the 8th, 17th, and 25th/final week of postnatal intervention curriculum. (Baseline & approx. 2, 4, 6 & 8 mos from each peer group's start, respectively.)
  Breastfeeding intent, initiation, and duration will be assessed using a survey
Introduction of solid foods and sugar-sweetened beverages | After (within 31 days of) the 25th/final week of the postnatal intervention curriculum. (Approximately 8 months from each peer group's start.)
  Timing of initiation of solid foods and sugar sweetened beverages will be assessed using a survey.
Infant sleep behaviors | At (or within 31 days of) the infant's newborn primary care visit, and during (or within 31 days of ) the 8th, 17th, and 25th/final week of the postnatal intervention curriculum. (Approx. 2, 4, 6 and 8 months from each peer group's start, respectively.)
  Infant sleeping and related maternal activities will be measured using the validated Brief Infant Sleep Questionnaire (BISQ). Subjects will complete the abbreviated 13-item BISQ (A-BISQ), as well as 2 additional questions from the expanded version (E-BISQ).
Parenting self-efficacy | At (or within 31 days of) the 8th and 25th/final weeks of the postnatal intervention curriculum. (Approx. 4 and 8 months from each peer group's start, respectively.)
  The Karitane Parenting Confidence Scale (KPCS) is a 15-item validated scale that will be used to measure parenting self-efficacy. Questions assess the frequency of certain beliefs, skills and abilities related to successful parenting, measured using a 4-point response structure (No, hardly ever; No, not very often; Yes, some of the time; Yes, most of the time).
Positive parenting behaviors | At (or within 31 days of) the infant's newborn primary care visit, and during (or within 31 days of ) the 8th and 25th/final week of the postnatal intervention curriculum. (Approx. 2, 4, and 8 months from each peer group's start, respectively).
  Mothers will be assessed regarding specific parenting practices using the 10-item Infant/Toddler (IT) Home Observation for Measurement of the Environment (HOME) Inventory. Individual responses for each yes/no item are coded to 0 or 1.
Maternal self-care behaviors | At (or within 31 days of) the infant's newborn primary care visit, and during (or within 31 days of ) the 8th, 17th, and 25th/final week of the postnatal intervention curriculum. (Approx. 2, 4, 6 and 8 months from each peer group's start, respectively.)
  Mothers will be asked 11 questions related to their self-care behaviors, including their own sleep habits, support-seeking behaviors, and taking time for themselves. These items are a combination of Likert-scaled items and simple measures of the frequency of behaviors.
Maternal social support | At enrollment and during (within 31 days of) the 25th/final week of the postnatal intervention curriculum. (Baseline & approximately 8 mos from each peer group's start, respectively.)
  Mothers' level of social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS). This validated scale is made up of 12 items. Responses for this scale are coded from 1 to 7 (very strongly disagree, strongly disagree, mildly disagree, neutral, mildly agree, strongly agree, and very strongly agree).
Maternal depression | At (or within 31 days of) the 8th and 25th/final weeks of the postnatal intervention curriculum. (Approx. 4 and 8 months from each peer group's start, respectively.)
  The Patient Health Questionnaire-9 (PHQ-9), a validated 9-item scale, will be used to measure maternal depression at follow-up visits. This brief scale asks about the frequency of depression symptoms experienced over the past week (where 0 = Not at all, 1 = Several days, 2 = More than half the days, and 3 = Nearly every day), and produces an overall score ranging from 0 - 27. Participants who score 10 or greater will be contacted, screened for suicidality by a psychologist and offered referrals to supportive services.
Maternal stress | At (or within 31 days of) the 8th and 25th/final weeks of the postnatal intervention curriculum. (Approx. 4 and 8 months from each peer group's start, respectively.)
  The Parental Stress Scale (PSS) is a validated, 18-item public domain scale measuring perceived parental stress using a 5-point Likert rating scale ('Strongly disagree' to 'strongly agree').
Infant weight and growth | At (or within 31 days of) the 8th and 25th/final weeks of the postnatal intervention curriculum. (Approx. 4 and 8 months from each peer group's start, respectively.)
  Infants' weight will be measured using a calibrated digital scale and length will be measured using a standard infantometer. Measurements will be taken by a member of the study staff trained in anthropometric measures. Infants birth weight will also be obtained from medical records.
Contraceptive use: Intent and behaviors | At enrollment, and after (within 31 days of) the 25th/final week of the postnatal intervention curriculum (approximately 8 months from each peer group's start.)
  At enrollment, future plans for contraceptive use will be assessed; in the final survey, 3 questionnaire items will assess contraceptive use behaviors since delivery. All questionnaire items have been adapted from the Centers for Disease Control and Prevention (CDC) Youth Risk Behavior Survey (YRBS).
Maternal weight and height | At (or within 31 days of) the 8th and 25th/final weeks of the postnatal intervention curriculum. (Approx. 4 and 8 months from each peer group's start, respectively.)
  Mothers' weight will be measured using a calibrated digital scale and height will be measured using a standard stadiometer. Measurements will be taken by a member of the study staff trained in anthropometric measures. Maternal pre-pregnancy height and weight will also be obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G. Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania